CLINICAL TRIAL: NCT03246776
Title: The Clinical Study of the Microbial Colonization of Chronic Keratinized Hand Eczema and the Change of Microbial Colonization After External Using of Halometasone Triclosan Cream
Brief Title: Microbial Colonization and Change of Chronic Keratinized Hand Eczema After Using Halometasone Triclosan
Acronym: MCCK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Wei Xu, associated professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BeijingFH20170801
Record Dates: First submitted 2017-08-02; First posted 2017-08-11 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Chronic Hand Eczema

STUDY DESIGN:
Masking Description: open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Halometasone Triclosan Cream (Experimental): All subjects receive external Use of Halometasone Triclosan Cream
  Interventions: Drug: Halometasone Triclosan

INTERVENTIONS:
Drug: Halometasone Triclosan — Halometasone Triclosan . The study product will be applied topically twice a day (morning and evening) for 14 days of treatment
  Other Names: regular moisturizer; wet wrap bandage

SUMMARY:
The clinical study of the microbial colonization of chronic keratinized hand eczema and the change of microbial colonization after external using of Halometasone Triclosan Cream

DETAILED DESCRIPTION:
The clinical study of the microbial colonization of chronic keratinized hand eczema and the change of microbial colonization after external using of Halometasone Triclosan Cream

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Chronic Keratinized hand eczema for at least 3 months
* The affected area is greater than 30%
* Overall assessment of the severity of the disease(IGA)≥3 OR HEES≥13
* No obvious incentive .Who have read the instructions of the subject, agreed to and signed written informed consent, and have been able to provide a personal medical history.

Exclusion Criteria:

* Pregnancy, breast feeding
* Severe liver and kidney disease, blood system disease, autoimmune disease, chronic severe infection, diabetes, mental illness, drug use, alcohol abuse, etc
* Malignant neoplasms or other serious maladies that may affect the correct assessment of efficacy
* Topical corticosteroid was suspended for less than 2 weeks;The system used corticosteroids and other immunosuppressive agents (thunder vine and other drugs) which were suspended for less than four weeks
* Eczema of the facial and skin creases
* Atopic dermatitis, contact dermatitis, blister hand eczema, contact urticaria, discoid eczema
* participated in other clinical trials within 3 months.
* Known sensitivity to Halometasone Triclosan
* failure to follow the prescribed medication or the incomplete record of the test process which will affect the curative effect judgment
* Other reasons why researchers think they should not be included

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-08-20 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Response to Hand eczema severity | 2 weeks
  HEES(hand eczema extent score)

SECONDARY OUTCOMES:
Response to treatment/Hand eczema severity | 2 weeks
  Photographic evaluation
Investigator reported improvement | 2 weeks
  IGA(investigator's global assessment)
Response to treatment/Hand eczema severity | 2 weeks
  Dermatoscopy
Response to Quality of Life | week 0 and 2
  questionnaire :DLQI(dermatology life quality index)
Patient Reported Improvement | up to 2 weeks
  VAS(Visual Analog Score for pruritus)
Response to treatment/Hand eczema severity | 2 weeks
  HECSI
Response to Microbial Colonization rates | 2 weeks
  Staphylococcus aureus colonization rates

CONTACTS AND LOCATIONS:
Overall Officials: linfeng li, phd, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided